CLINICAL TRIAL: NCT00748384
Title: Usability of the Foresee Home in Intermediate Age Related Macular Degeneration Patients
Brief Title: Usability of the Foresee Home in Intermediate Age Related Macular Degeneration (AMD) Patients
Acronym: UU2
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: HMP-UU2
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Age Related Macular Degeneration
Keywords: HMP, CNV, AMD, PHP, HPHP, foresee
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Self trained subjects
- 2: supervised trained subjects

SUMMARY:
The study purpose is to demonstrate that the target population can receive a packed FORESEE HOME unpack it, install and operate it to an extent that the FORESEE HOME can monitor them for changes in the visual field with good specificity. And evaluate the device usage on a small scale, at the subjects' homes before a commercial use.

DETAILED DESCRIPTION:
Numerical output of the FORESEE HOME, output of the usability parameters provided by the FORESEE HOME device, counts of the number of subjects who successfully set up the device and conduct testing sessions.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to sign a consent form and participate in the study

  * Subjects diagnosed as intermediate AMD in at least one eye (in case a patient will convert during the study period he will be excluded)
  * Age more than 50 years
  * VA with habitual correction better than 20/60 in the study eye
  * Ability to speak, read and understand instructions in English or Hebrew
  * Familiar with computer usage

Exclusion Criteria:

* Evidence of macular disease other than AMD or glaucoma in the study eye

  * Presence of any significant media opacity that precludes a clear view of the macular area as identified in the study eye by biomicroscopy, CFP.
  * Any non-macular related ocular surgery performed within 3 months prior to study entry in the target eye
  * Never been tested on the PHP device
  * Participation in another study with the exclusion of AREDS study
  * Patients diagnosed with geographic atrophy (GA)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed as Intermediate AMD
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who managed to set the device | 6 months
Proportion of subjects who managed to perform the test after dynamic tutorial/supervised training | 6 month
Number of device malfunctions | 6 month
Average use of the device | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Haya Morori Katz, M.D., Principal Investigator — Kaplan Medical Center
Locations (2):
- Israel (2):
  - Meir Medical Center, Kfar Saba
  - Kaplan Medical Center, Rehovot

REFERENCES:
- See also: sponsor site — http://www.notalvision.com